CLINICAL TRIAL: NCT01145924
Title: Transbronchial Needle Forceps for EBUS
Brief Title: Transbronchial Needle Forceps for Endobronchial Ultrasound
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Prof. Felix JF Herth, Thoraxklinik Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HD 08
Record Dates: First submitted 2010-06-07; First posted 2010-06-17 (Estimated); Last update posted 2010-06-17 (Estimated); Status verified 2010-02

CONDITIONS: Lung Cancer; Lymph Nodes
Keywords: bronchoscopy; endobronchial ultrasound; transbronchial needle aspiration; lung cancer; staging
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EBUS TBNF (Active Comparator): single arm trial, patients with enlarged mediastinal nodes will be examine
  Interventions: Procedure: EBUS TBNF

INTERVENTIONS:
Procedure: EBUS TBNF — Transbronchial needle forceps will be use with the EBUS TBNA scope
  Other Names: Endobronchial ultrasound

SUMMARY:
Prove the feasibility of a needle forceps in patients with enlarged mediastinal lymph nodes

DETAILED DESCRIPTION:
Patients with enlarged mediastinal lymph nodes must be staged. The EBUS TBNA technique is an established technique. Unfortunately the size of the needle is limited to 21 gauge. With tne new designed needle forceps it should be possible to obtain more material and establish the diagnosis more often

ELIGIBILITY:
Inclusion Criteria:

* enlarged mediastinal lymph nodes

Exclusion Criteria:

* comorbidities

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-08 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a positive biopsy result | 2 days after intervention

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 3 weeks after

CONTACTS AND LOCATIONS:
Overall Officials: Hendrik Dienemann, PhD, MD, Study Director — Heidelberg University
Locations (1):
- Thoraxklinik, Heidelberg, Germany

REFERENCES:
- [Derived] Herth FJ, Schuler H, Gompelmann D, Kahn N, Gasparini S, Ernst A, Schuhmann M, Eberhardt R. Endobronchial ultrasound-guided lymph node biopsy with transbronchial needle forceps: a pilot study. Eur Respir J. 2012 Feb;39(2):373-7. doi: 10.1183/09031936.00033311. Epub 2011 Jun 23. PMID 21700609